CLINICAL TRIAL: NCT02766179
Title: A Randomized Cross-over Study of Adjustable Thermoplastic Oral Appliances and Continuous Positive Airway Pressure in Treatment of Patients With Obstructive Sleep Apnea
Brief Title: Compare Outcomes of SMG and CPAP in OSA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, WISH BANHIRAN, Associate Professor, Mahidol University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: R015733017
Record Dates: First submitted 2016-05-04; First posted 2016-05-09 (Estimated); Last update posted 2016-05-09 (Estimated); Status verified 2016-05

CONDITIONS: Quality of Life; Sleep Apnea Syndromes
MeSH Terms: conditions — Sleep Apnea Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CPAP Therapy (Active Comparator): Continuous Positive Airway Pressure
  Interventions: Device: CPAP
- Somnoguard (Experimental): Somnoguard
  Interventions: Device: Somnoguard

INTERVENTIONS:
Device: CPAP — CPAP is used for 6 weeks
  Other Names: Continuous positive airway pressure therapy
  Arms: CPAP Therapy
Device: Somnoguard — Somnoguard is used for 6 weeks
  Arms: Somnoguard

SUMMARY:
The objectives of this study is to compare short-term outcomes of CPAP and Adjustable thermoplastic oral appliance in the treatment of obstructive sleep apnea. Study design is a randomized cross-over trial during 6-week period of each treatment in 50 patients. Primary outcomes are quality of life, degree of sleepiness, and severity of OSA determined by FOSQ ESS, and AHI or RDI, respectively.

DETAILED DESCRIPTION:
The objectives of this study is to compare short-term outcomes of CPAP and Adjustable thermoplastic oral appliance in the treatment of obstructive sleep apnea. Study design is a randomized cross-over trial during 6-week period of each treatment in 50 patients. Primary outcomes are quality of life, degree of sleepiness, and severity of OSA determined by FOSQ ESS, and AHI or RDI, respectively. Wash-in period 2 weeks and Wash-out periods 2 weeks are required before start each treatment.

ELIGIBILITY:
Inclusion Criteria:

1. OSA patients aged over 18 YO at Siriraj hospital
2. AHI 5 - 30 events/ h or AHI > 30 events/h but lowest O2 saturation > 70%
3. Positive consented form

Exclusion Criteria:

1. Patients with severe Temporomandibular joint diseases or limited mandible advancement (< 5 mm)
2. Patients with severe periodontal diseases or inadequate teeth (< 3 teeth in each quadrant)
3. Patients with unstable medical problems i.e. poorly controlled cardiovascular diseases, COPD, cancers, cerebrovascular diseases, epilepsy, dementia, etc.
4. Patients who could not tolerate the side effects of CPAP or SMG
5. Patients who could not follow-up until finishing the protocol or withdraw themselves from the study for any reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2014-10; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Quality of life | 6 weeks
  FOSQ scores

SECONDARY OUTCOMES:
side effects | 6 weeks
  questionnaires
satisfaction | 6 weeks
  VAS scores
AHI | 6 weeks
  Apnea-hypopnea index (events per hour)
Degree of sleepiness | 6 weeks
  ESS scores
lowest oxygen saturation | 6 weeks
  lowest oxygen saturation (%)

CONTACTS AND LOCATIONS:
Overall Officials: Wish Banhiran, MD, Principal Investigator — Siriraj Hospital
Locations (1):
- Siriraj Hospital, Bangkok, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Banhiran W, Assanasen P, Nopmaneejumrudlers C, Nujchanart N, Srechareon W, Chongkolwatana C, Metheetrairut C. Adjustable thermoplastic oral appliance versus positive airway pressure for obstructive sleep apnea. Laryngoscope. 2018 Feb;128(2):516-522. doi: 10.1002/lary.26753. Epub 2017 Jul 17. PMID 28714534